CLINICAL TRIAL: NCT01664507
Title: The Effect and Safety of Low Dose Nebulized Epinephrine in the Treatment of Croup
Brief Title: The Effect and Safety of Low Dose Nebulized Epinephrine in Croup
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Hee Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Croup_01
Record Dates: First submitted 2012-08-03; First posted 2012-08-14 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Croup; Epinephrine, Administration, Inhalation
Keywords: croup, dose, epinephrine
MeSH Terms: conditions — Croup; Respiratory Aspiration | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional dose epinephrine (Active Comparator): L-epinephrine (1:1000) 0.5 mL/kg (maximum 5mL) + normal saline : total 5mL
  Interventions: Drug: conventional dose epinephrine
- low dose epinephrine (Experimental): L-epinephrine (1:1000) 0.1 mL/kg (maximum 1mL) + normal saline : total 5mL
  Interventions: Drug: low dose epinephrine

INTERVENTIONS:
Drug: conventional dose epinephrine — conventional dose epinephrine : 0.5mg/kg + 0.9% normal saline
  Arms: conventional dose epinephrine
Drug: low dose epinephrine — low dose epineprhine : 0.1mg/kg + 0.9% normal saline
  Arms: low dose epinephrine

SUMMARY:
Croup is common illness presenting emergency department with dyspnea. The main treatment for croup is nebulized L-epinephrine and steroid. The study for the dose of nebulized L-epinephrine is restricted that the study of comparision between racemic epinephrine and L-epinephrine.

The investigators conducted this study to compare the effectiveness of low dose L-epinephrine with conventional dose L-epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* croup children between 6 month and 5 years old
* Westley croup score between 3 and 11

Exclusion Criteria:

* underlying lung or heart disase
* contra indication to dexamethasone
* immune deficient state
* preterm birth
* previous intubation or apnea history

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
the difference of Westley croup score between baseline and 30 minutes after neublized treatment | 30 minutes

SECONDARY OUTCOMES:
the incidence of use of additional neublized treatment | 30 minutes
Westley croup score | 30, 60, 90, 120, 180, 240 minutes
the side effect of epinephrine | participants will be followed for the duration of ED stay
  Hypertension, tachycardia : more than 95th percentile for age Arrythmia Pallor Tremor
respiratory rate, oxygen saturation | 30, 60, 90, 120, 180, 240 minutes
health care utilization- length of stay in emergency department, admission rate, revisit dut to croup symptom | within 7 days
treatment failure | 30min after 2nd epinephrine nebulizer
  after additional nebulized epineprhine at 30 minutes, as the croup scrore is higher than baselin, the blinding is cleared.
rebound effect | 180 minutes
  the croup score is the same or over than the base line

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Jung JY, Lee HJ, Kim DK, Kwak YH, Chang I, Kwon H, Choi YJ, Park JW, Paek SH, Cho JH. Efficacy of low-dose nebulized epinephrine as treatment for croup: A randomized, placebo-controlled, double-blind trial. Am J Emerg Med. 2019 Dec;37(12):2171-2176. doi: 10.1016/j.ajem.2019.03.012. Epub 2019 Mar 8. PMID 30878411